CLINICAL TRIAL: NCT06373614
Title: The Effect of Foot Massage and Bed Bath on Fatigue and Sleep Quality in Individuals With Cancer.
Brief Title: The Effect of Foot Massage and Bed Bath on Individuals With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/18
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Patients
Keywords: cancer; sleep quality; fatigue; bed bath; foot massage
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: foot massage (intervention group) bed bath (intervention group) control (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- foot massage (Experimental): Foot massage will be applied for a total of 30 minutes, 15 on the right foot and 15 on the left foot. In order to move comfortably during the foot massage, non-allergenic baby oil will be used. This intervention will continue in the evenings for 4 days.
  Interventions: Other: foot massage
- bed bath (Experimental): Bed bath will be applied for a total of 30 minutes with cotton and warm water. This intervention will continue in the evenings for 4 days.
  Interventions: Other: bed bath
- control (No Intervention): no intervention

INTERVENTIONS:
Other: foot massage — Interventions are to be performed in the evening before bedtime for 4 consecutive days.
  Arms: foot massage
Other: bed bath — Interventions are to be performed in the evening before bedtime for 4 consecutive days.
  Arms: bed bath

SUMMARY:
Foot massage or bed bath will be applied to improve sleep quality and reduce fatigue levels of individuals with cancer.

DETAILED DESCRIPTION:
Foot massage provides relaxation of the body with rubbing movements applied to the feet. The bathroom was an important part of the individual's general hygienic care In addition, it also ensures the physical and psychological comfort, safety and well-being of the individual.Massage and bed bath are among the independent interventions of the nurse that help the individual to relax within the scope of the Nursing Regulation. This study was planned to determine the effect of foot massage and bed bath on fatigue and sleep level in individuals with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* illiterate,
* diagnosed with cancer
* volunteer to participate in the study

Exclusion Criteria:

* unable to communicate verbally
* Patients who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
sleep quality | In the study, the sleep quality of the patients will be evaluated for 5 days after the sleep.
  The effect of interventions on sleep will be measured. The Richard Cample Sleep Scale will be used for this. A score of "0-25" indicates "very poor sleep" and a score of "76-100" indicates "very good sleep".
fatigue | In the study, the fatigue of the patients will be evaluated for 5 days in the evening, before the interventions.
  The effect of interventions on fatigue will be measured. Brief Fatigue Invantory; (BFI) will be used for this. Scoring the items are between "0" and "10", where "0" means not affected at all and "10" means affected at the highest level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ı want to share my research protocol after the publication.

REFERENCES:
- [Background] Mazloum SR, Rajabzadeh M, Mohajer S, Bahrami-Taghanaki H, Namazinia M. Comparing the Effects of Warm Footbath and Foot Reflexology on the Fatigue of Patients Undergoing Radiotherapy: A Randomized Clinical Trial. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231172940. doi: 10.1177/15347354231172940. PMID 37162156
- [Result] Richards K. Techniques for measurement of sleep in critical care. Focus Crit Care. 1987 Aug;14(4):34-40. No abstract available. PMID 3650169
- [Result] Schoonhoven L, van Gaal BG, Teerenstra S, Adang E, van der Vleuten C, van Achterberg T. Cost-consequence analysis of "washing without water" for nursing home residents: a cluster randomized trial. Int J Nurs Stud. 2015 Jan;52(1):112-20. doi: 10.1016/j.ijnurstu.2014.08.001. Epub 2014 Aug 10. PMID 25173772
- [Result] Quattrin R, Zanini A, Buchini S, Turello D, Annunziata MA, Vidotti C, Colombatti A, Brusaferro S. Use of reflexology foot massage to reduce anxiety in hospitalized cancer patients in chemotherapy treatment: methodology and outcomes. J Nurs Manag. 2006 Mar;14(2):96-105. doi: 10.1111/j.1365-2934.2006.00557.x. PMID 16487421
- [Derived] Kabuk A, Demirel U, Inangil D. The effectiveness of nursing interventions on fatigue and sleep quality in hospitalized cancer patients: the role of foot massage and bed bath. Support Care Cancer. 2026 Feb 5;34(3):169. doi: 10.1007/s00520-026-10386-7. PMID 41644843